CLINICAL TRIAL: NCT03038672
Title: A Randomized Phase 2 Study of CDX-1127 (Varlilumab) in Combination With Nivolumab in Patients With Relapsed or Refractory Aggressive B-cell Lymphomas
Brief Title: Nivolumab With or Without Varlilumab in Treating Patients With Relapsed or Refractory Aggressive B-cell Lymphomas
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-00120; NCI-2017-00120 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC168D; 10089 (Other: Dana-Farber - Harvard Cancer Center LAO); 10089 (Other: CTEP); UM1CA186686 (NIH); UM1CA186709 (NIH)
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Results first posted 2024-10-16 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: ALK-Positive Large B-Cell Lymphoma; Diffuse Large B-Cell Lymphoma Activated B-Cell Type; Diffuse Large B-Cell Lymphoma Associated With Chronic Inflammation; Diffuse Large B-Cell Lymphoma Germinal Center B-Cell Type; Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; EBV-Positive Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; EBV-Positive Mucocutaneous Ulcer; HHV8-Positive Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; High Grade B-Cell Lymphoma With MYC and BCL2 and/or BCL6 Rearrangements; High Grade B-Cell Lymphoma, Not Otherwise Specified; Intravascular Large B-Cell Lymphoma; Large B-Cell Lymphoma With 11q Aberration; Large B-Cell Lymphoma With IRF4 Rearrangement; Plasmablastic Lymphoma; Primary Diffuse Large B-Cell Lymphoma of the Central Nervous System; Primary Effusion Lymphoma; Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Burkitt Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Gray-Zone Lymphoma; Recurrent High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Recurrent High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; Recurrent Lymphomatoid Granulomatosis; Recurrent Primary Cutaneous Diffuse Large B-Cell Lymphoma, Leg Type; Recurrent Primary Mediastinal Large B-Cell Lymphoma; Recurrent T-Cell/Histiocyte-Rich Large B-Cell Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Burkitt Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Gray-Zone Lymphoma; Refractory High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Refractory High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; Refractory Primary Cutaneous Diffuse Large B-Cell Lymphoma, Leg Type; Refractory Primary Mediastinal Large B-Cell Lymphoma; Refractory T-Cell/Histiocyte-Rich Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Plasmablastic Lymphoma; Lymphoma, Primary Effusion; Lymphoma, B-Cell; Burkitt Lymphoma; Lymphomatoid Granulomatosis | interventions — Nivolumab; varlilumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (nivolumab) (Active Comparator): Patients receive nivolumab IV over 30 minutes every 2 weeks for 4 months and every 4 weeks for a total of up to 2 years in the absence of disease progression or unacceptable toxicity. Patients may cross over to Group II at the time of disease progression.
  Interventions: Biological: Nivolumab
- Group II (varlilumab, nivolumab) (Experimental): Patients receive varlilumab IV over 90 minutes every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also receive nivolumab IV over 30 minutes every 2 weeks for 4 months and every 4 weeks for a total of up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab; Drug: Varlilumab

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Drug: Varlilumab — Given IV
  Other Names: CDX 1127; CDX-1127; CDX1127; Immunoglobulin G1, Anti-(Human CD Antigen CD27) (Human Monoclonal CDX-1127 Clone 1f5 Heavy Chain), Disulfide with Human Monoclonal CDX-1127 Clone 1f5 Kappa-chain, Dimer
  Arms: Group II (varlilumab, nivolumab)

SUMMARY:
This phase II trial studies how well nivolumab with or without varlilumab works in treating patients with aggressive B-cell lymphomas that have come back (recurrent) or do not respond to treatment (refractory). Immunotherapy with monoclonal antibodies, such as varlilumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the anti-tumor activity of combination therapy with CDX-1127 (varlilumab) and nivolumab as compared to nivolumab alone in patients with advanced aggressive B-cell non-Hodgkin lymphomas (NHL) based on the lymphoma response to immunomodulatory therapy criteria or LYRIC.

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability profile of treatment with a combination of CDX-1127 (varlilumab) and nivolumab in patients with advanced aggressive B-cell NHL.

II. To evaluate the duration of response, progression-free survival and overall survival.

EXPLORATORY OBJECTIVES:

I. To determine the effect of combination therapy with CDX-1127 (varlilumab) and nivolumab on the immune system as assessed by immunohistochemistry (IHC), mass cytometry (CyTOF), changes in serum cytokine profile and immunogenicity assays.

II. To describe the pharmacokinetic profile of CDX-1127 (varlilumab) and nivolumab when used in combination.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive nivolumab intravenously (IV) over 30 minutes every 2 weeks for 4 months and every 4 weeks for a total of up to 2 years in the absence of disease progression or unacceptable toxicity. Patients may cross over to Group II at the time of disease progression.

GROUP II: Patients receive varlilumab IV over 90 minutes every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also receive nivolumab IV over 30 minutes every 2 weeks for 4 months and every 4 weeks for a total of up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 100 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histopathologically confirmed diagnosis of an aggressive B-cell non-Hodgkin lymphoma that is recurrent or refractory to standard therapy
* For the purpose of this study, aggressive B-cell NHL will be deemed any lymphoma belonging to one of the following groups according to the 2016 revision of the World Health Organization (WHO) classification of lymphoid neoplasms

  * For the purposes of stratification, diagnoses are grouped into 2 categories:

    * Category A

      * Burkitt lymphoma
      * Burkitt-like lymphoma with 11q aberration
      * High-grade B-cell lymphoma, with MYC and BCL2 and/or BCL6 rearrangements
      * High-grade B-cell lymphoma, not otherwise specified (NOS)
    * Category B

      * Diffuse large B-cell lymphoma (DLBCL), NOS
      * Diffuse large B-cell lymphoma (DLBCL), NOS; germinal center B-cell type
      * Diffuse large B-cell lymphoma (DLBCL), NOS; activated B-cell type
      * Large B-cell lymphoma with IRF4 rearrangement
      * T-cell/histiocyte-rich large B-cell lymphoma
      * Primary DLBCL of the central nervous system (CNS)
      * Primary cutaneous DLBCL, leg type
      * Epstein-Barr virus (EBV)+ DLBCL, NOS
      * EBV+ mucocutaneous ulcer
      * DLBCL associated with chronic inflammation
      * Lymphomatoid granulomatosis
      * Primary mediastinal (thymic) large B-cell lymphoma
      * Intravascular large B-cell lymphoma
      * ALK+ large B-cell lymphoma
      * Plasmablastic lymphoma
      * Primary effusion lymphoma
      * Human herpesvirus (HHV)-8+ DLBCL, NOS
      * B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and classical Hodgkin lymphoma
* Patients must have measurable disease, defined as at least one lesion that is > 15 mm (1.5 cm) in the longest axis on cross-sectional imaging and measurable in two perpendicular dimensions per computed tomography (spiral computed tomography [CT]), positron emission tomography (PET)-CT or magnetic resonance imaging (MRI)
* Patients must have disease that has relapsed after or is refractory to at least 2 lines of standard therapy; the remaining standard treatment options are unlikely to be effective in the opinion of the treating physician, or patient is felt to be ineligible for such therapies or the patient refuses such therapies; patients who have undergone autologous stem cell transplant are eligible as long as they meet all other criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of greater than 12 weeks
* White blood cell (WBC) >= 2000/mm^3 (within 14 days of registration)
* Absolute neutrophil count (ANC) >= 1500/mm^3 (within 14 days of registration)
* Platelet count >= 100,000/mm^3 (within 14 days of registration)
* Hemoglobin > 9.0 g/dL (within 14 days of registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (except patients with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL) (within 14 days of registration)
* Aspartate transaminase (aspartate aminotransferase [AST]) =< 2.5 x ULN (within 14 days of registration)
* Calculated creatinine clearance (CrCl) >= 50 mL/min (if using the Cockcroft-Gault formula) (within 14 days of registration)
* Females of child bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG])
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patient has received chemotherapy, targeted agent, or radiotherapy within 4 weeks or at least 5 half-lives, whichever is longer, prior to registration
* Palliative (limited-field) radiation therapy is permitted, if all of the following criteria are met:

  * Repeat imaging demonstrates no new sites of bone metastases
  * The lesion being considered for palliative radiation is not a target lesion
* Patient has received immunotherapy (including monoclonal antibodies) within 4 weeks prior to registration
* Patients who have not recovered to grade 1 or less from any adverse events due to agents administered more than 4 weeks earlier (excluding alopecia)
* Patients who are receiving any other investigational agents
* Patients should be excluded if they have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Patients who have received autologous stem cell transplant (ASCT) =< 12 weeks prior to the first dose of study drug
* Patients with a prior history of allogeneic stem cell or solid organ transplantation
* Patients with evidence of active disease in the central nervous system (CNS) defined as either the presence of active lesions on MRI obtained within 4 weeks of registration or progressive neurological decline

  * Patients with primary CNS lymphoma who develop systemic recurrence following standard therapy may be included as long as no active CNS disease is present at the time or enrollment; similarly, patients with secondary involvement of the CNS from a systemic lymphoma may be included as long as the CNS disease has been optimally treated and they demonstrate no evidence of active CNS disease
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CDX-1127 (varlilumab) and/or nivolumab
* History of severe hypersensitivity reaction to any monoclonal antibody
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because CDX-1127 (varlilumab) and nivolumab are agents with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CDX-1127 (varlilumab) or nivolumab, breastfeeding should be discontinued if the mother is treated with CDX-1127 (varlilumab) or nivolumab
* Patients with human immunodeficiency virus (HIV) are eligible for the study provided they meet the other protocol criteria in addition to the following:

  * Undetectable HIV load by standard polymerase chain reaction (PCR) clinical assay within 60 days prior to registration
  * Absolute CD4 count of >= 200 mm^3 within 60 days prior to registration
  * Willing to maintain adherence to combination antiretroviral therapy
  * No history of acquired immunodeficiency syndrome (AIDS) defining condition (other than lymphoma or CD4 cell count < 200 mm^3)
  * Likely to have near normal lifespan if not for the presence of relapsed/refractory lymphoma

    * Patients with evidence of hepatitis B virus (HBV) are eligible provided there is minimal hepatic injury and the patient has undetectable HBV on suppressive HBV therapy; patient must be willing to maintain adherence to HBV therapy
    * Patients with previously treated and eradicated hepatitis C virus (HCV) who have minimal hepatic injury are eligible
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded; these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease; patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible; patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption); physiologic replacement doses of systemic corticosteroids are permitted, even if =< 10 mg/day prednisone equivalents; a brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study
* Patients with other active malignancy =< 3 years prior to registration for which active treatment is required must be excluded; patients with composite lymphomas that have a non-B-cell component must be excluded EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2026-10-24 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Ansell, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (33):
- United States (33):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Period: Initial Treatment
Arm/Group | Group I (Nivolumab) | Group II (Varlilumab, Nivolumab)
Started | 27 | 27
Completed | 25 | 26
Not Completed | 2 | 1
Not completed — Unacceptable chemistry | 0 | 1
Not completed — Progression prior to treatment | 1 | 0
Not completed — No treatment per protocol | 1 | 0
Period: Cross Over From Group I to Group II
Arm/Group | Group I (Nivolumab) | Group II (Varlilumab, Nivolumab)
Started | 7 | 26
Completed | 7 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Nivolumab) | Group II (Varlilumab, Nivolumab) | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Median (Full Range); unit: years] | 67 [21 to 84] | 69 [29 to 86] | 67.5 [21 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 19 | 20 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 27 | 24 | 51
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 24 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Will be assessed by computed tomography (CT)-based criteria or positron emission tomography (PET)-CT based criteria. A response will be defined as an objective status of partial remission (PR) or complete remission (CR) for patients evaluated by CT-based criteria and complete metabolic response (CMR) or partial metabolic response (PMR) for patients evaluated by PET-CT based criteria. Exact binomial ninety-five percent confidence intervals for the true success proportion will be calculated in each arm. Comparison of overall response rates between the two treatment groups will be performed using a one-sided Fisher's exact test at significance level 0.15.
Time Frame: 2 years
Population: All eligible patients that had a disease evaluation after being treated.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Group I (Nivolumab) | Group II (Varlilumab, Nivolumab)
Number analyzed (Participants) | 25 | 26
proportion of participants | 0.16 [0.045 to 0.361] | 0.08 [0.010 to 0.251]

2. Secondary Outcome: Duration of Response
Description: Defined as the date at which the patient's objective status is first noted to be a PR or CR for patients evaluated by CT-based criteria or CMR or PMR for patients evaluated by PET-CT based criteria to the earliest date progression (documentation of disease progression [PMD] or progressive disease [PD]) is documented. The distribution of duration of response will be estimated using the method of Kaplan-Meier. The comparison of duration of response between two treatment arms will be based on the log-rank test.
Time Frame: 2 years
Population: All eligible and treated patients that achieve a response.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Group I (Nivolumab) | Group II (Varlilumab, Nivolumab)
Number analyzed (Participants) | 4 | 2
years | NA [NA to NA] — Due to a lack of events the median and confidence intervals cannot be determined. | 0.2 [0.2 to NA] — Due to a lack of events the upper confidence interval cannot be determined.

3. Secondary Outcome: Overall Survival
Description: The distribution of survival time will be estimated using the method of Kaplan-Meier. The comparison of overall survival between two treatment arms will be based on the log-rank test.
Time Frame: 37 months
Population: All eligible and treated patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group I (Nivolumab) | Group II (Varlilumab, Nivolumab)
Number analyzed (Participants) | 25 | 26
Months | 8.6 [4.7 to NA] — Due to a lack of events the upper limit was not reached. | 10.2 [3.1 to NA] — Due to a lack of events the upper limit was not reached.

4. Secondary Outcome: Progression Free Survival (PFS)
Description: The distribution of PFS will be estimated using the method of Kaplan-Meier. The comparison of progression-free survival between two treatment arms will be based on the log-rank test.
Time Frame: 37 months
Population: All eligible and treated patients that had a disease evaluation.
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Group I (Nivolumab) | Group II (Varlilumab, Nivolumab)
Number analyzed (Participants) | 25 | 24
Months | 2.6 [1.5 to 3.2] | 1.5 [1.1 to 3.2]

5. Secondary Outcome: Proportion of Patients With Grade 3 or Higher Adverse Events
Description: Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The overall adverse event rates for grade 3 or higher hematologic and non-hematologic adverse events at least possibly related to treatment will be compared between the two treatment groups using the Chi-square test (or Fisher's exact test if the data in the contingency table is sparse).
Time Frame: 25 months
Population: All eligible and treated patients.
Measure: Number; unit: proportion of patients
Arm/Group | Group I (Nivolumab) | Group II (Varlilumab, Nivolumab)
Number analyzed (Participants) | 25 | 26
proportion of patients | 0.76 | 0.84

6. Other Pre Specified Outcome: Change in CD27 Expression in Tissue
Description: Will be assessed by immunohistochemistry. Will be both graphically and quantitatively summarized and explored. Standard paired comparisons methodologies (Wilcoxon signed rank and McNemar's tests) will be used to assess changes in these variables before and after therapy. In addition, baseline values and changes over time in each measure will be explored in relation to clinical outcome. Differences between responders and non-responders will be assessed using Wilcoxon's rank sum (continuous data) or Fisher's exact (categorical data) test. The relationship between each measure and time to event measures (PFS, overall survival [OS]) will be evaluated using Cox's proportional hazards models and log-rank tests. Logistic regression will be used to model the response rate as a function of treatment and CD27 (as a continuous variable). The distribution of CD27 will be estimated empirically in the entire trial population and used to calculate CD27 values corresponding to each fixed percentile.
Time Frame: Baseline up to 100 days after last dose of study drug
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Peripheral Blood Immune Cells
Description: Will be assessed by cytometry by time of flight (CyTOF). The relationship between presence/absence of a particular subtype of cell and association with outcomes will be evaluated. Evaluation of particular combinations of immune cells (immune signature) and whether they are predictive of outcome will also be evaluated. Will be both graphically and quantitatively summarized and explored. Standard paired comparisons methodologies (Wilcoxon signed rank and McNemar's tests) will be used to assess changes in these variables before and after therapy. In addition, baseline values and changes over time in each measure will be explored in relation to clinical outcome. Differences between responders and non-responders will be assessed using Wilcoxon's rank sum (continuous data) or Fisher's exact (categorical data) test. The relationship between each measure and time to event measures (PFS, OS) will be evaluated using Cox's proportional hazards models and log-rank tests.
Time Frame: Baseline up to 12 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in the Identification/Characterization of Intratumoral Immune Cells in Tissue
Description: Will be assessed by immunohistochemistry and CyTOF. Will be both graphically and quantitatively summarized and explored. Standard paired comparisons methodologies (Wilcoxon signed rank and McNemar's tests) will be used to assess changes in these variables before and after therapy. In addition, baseline values and changes over time in each measure will be explored in relation to clinical outcome. Differences between responders and non-responders will be assessed using Wilcoxon's rank sum (continuous data) or Fisher's exact (categorical data) test. The relationship between each measure and time to event measures (PFS, OS) will be evaluated using Cox's proportional hazards models and log-rank tests.
Time Frame: Baseline up to time of disease progression
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Genetic Alterations of Chromosome 9p24.1 in Tissue
Description: Will be assessed by fluorescence in situ hybridization. The proportion of patients in each of these groups who achieve a response will be evaluated. Will be both graphically and quantitatively summarized and explored. Standard paired comparisons methodologies (Wilcoxon signed rank and McNemar's tests) will be used to assess changes in these variables before and after therapy. In addition, baseline values and changes over time in each measure will be explored in relation to clinical outcome. Differences between responders and non-responders will be assessed using Wilcoxon's rank sum (continuous data) or Fisher's exact (categorical data) test. The relationship between each measure and time to event measures (PFS, OS) will be evaluated using Cox's proportional hazards models and log-rank tests.
Time Frame: Baseline up to time of disease progression
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Serum Cytokine Profile
Description: Will be assessed by enzyme-linked immunosorbent assay. Will be both graphically and quantitatively summarized and explored. Standard paired comparisons methodologies (Wilcoxon signed rank and McNemar's tests) will be used to assess changes in these variables before and after therapy. In addition, baseline values and changes over time in each measure will be explored in relation to clinical outcome. Differences between responders and non-responders will be assessed using Wilcoxon's rank sum (continuous data) or Fisher's exact (categorical data) test. The relationship between each measure and time to event measures (PFS, OS) will be evaluated using Cox's proportional hazards models and log-rank tests.
Time Frame: Baseline up to 12 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Mutation Burden in Tissue
Description: Will be assessed by whole exome sequencing. Will be both graphically and quantitatively summarized and explored. Standard paired comparisons methodologies (Wilcoxon signed rank and McNemar's tests) will be used to assess changes in these variables before and after therapy. In addition, baseline values and changes over time in each measure will be explored in relation to clinical outcome. Differences between responders and non-responders will be assessed using Wilcoxon's rank sum (continuous data) or Fisher's exact (categorical data) test. The relationship between each measure and time to event measures (PFS, OS) will be evaluated using Cox's proportional hazards models and log-rank tests.
Time Frame: Baseline up to time of disease progression
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 25 months for adverse events and 37 months for mortality
Groups:
- Cross Over to Group II Treatment (Varlilumab, Nivolumab): Pre cross over patients receive nivolumab IV over 30 minutes every 2 weeks for 4 months and every 4 weeks for a total of up to 2 years in the absence of disease progression or unacceptable toxicity. Patients may cross over to Group II at the time of disease progression.
  Post cross over patients receive varlilumab IV over 90 minutes every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also receive nivolumab IV over 30 minutes every 2 weeks for 4 months and every 4 weeks for a total of up to 2 years in the absence of disease progression or unacceptable toxicity.
Arm/Group | Group I (Nivolumab) | Group II (Varlilumab, Nivolumab) | Cross Over to Group II Treatment (Varlilumab, Nivolumab)
All-Cause Mortality (participants affected / at risk) | 3/27 | 5/27 | 0/7
Serious Adverse Events (participants affected / at risk) | 10/27 | 12/27 | 3/7
Other Adverse Events (participants affected / at risk) | 24/27 | 24/27 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Nivolumab) (N=27) | Group II (Varlilumab, Nivolumab) (N=27) | Cross Over to Group II Treatment (Varlilumab, Nivolumab) (N=7)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 2 (2) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (Nivolumab) (N=27) | Group II (Varlilumab, Nivolumab) (N=27) | Cross Over to Group II Treatment (Varlilumab, Nivolumab) (N=7)
Anemia (Blood and lymphatic system disorders) | 8 (8) | 13 (18) | 1 (1)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 3 (3) | 5 (5) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 4 (4) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 3 (4) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 6 (7) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (6) | 5 (5) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 6 (6) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 9 (11) | 3 (3)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 5 (5) | 3 (3)
Chills (General disorders) | 2 (2) | 2 (2) | 1 (1)
Edema limbs (General disorders) | 3 (3) | 4 (4) | 1 (1)
Fatigue (General disorders) | 9 (11) | 14 (18) | 2 (2)
Fever (General disorders) | 1 (1) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 4 (5) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 1 (2) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 3 (3) | 3 (4) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 4 (4) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Investigations - Other, specify (Investigations) | 2 (2) | 6 (6) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 9 (11) | 12 (16) | 6 (9)
Neutrophil count decreased (Investigations) | 2 (5) | 4 (8) | 0 (0)
Platelet count decreased (Investigations) | 4 (5) | 8 (14) | 0 (0)
Serum amylase increased (Investigations) | 2 (2) | 0 (0) | 1 (2)
Weight gain (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 1 (1) | 2 (2)
White blood cell decreased (Investigations) | 4 (7) | 6 (9) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 8 (11) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (5) | 4 (7) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5) | 7 (7) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 5 (7) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 4 (5) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) | 3 (3) | 2 (2)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 6 (7) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 2 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 4 (4) | 2 (2)
Lethargy (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 1 (1)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (3) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 4 (6) | 5 (5) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT03038672/Prot_SAP_000.pdf